CLINICAL TRIAL: NCT00911521
Title: Immunogenicity and Safety of a Quadrivalent Human Papillomavirus (HPV) Vaccine in Patients With Systemic Lupus Erythematosus (SLE): a Controlled Study
Brief Title: Immunogenicity and Safety of a Quadrivalent Human Papillomavirus (HPV) Vaccine in Patients With SLE: a Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NTWC/CREC/704/09
Record Dates: First submitted 2009-05-28; First posted 2009-06-02 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: human papillomavirus; vaccine; lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine arm (Active Comparator): subjects receiving vaccination
  Interventions: Drug: human papillomavirus vaccination (Gardasil)

INTERVENTIONS:
Drug: human papillomavirus vaccination (Gardasil) — 3 doses of the human papillomavirus vaccines to be given at baseline, month 2 and month 6
  Other Names: Gardasil

SUMMARY:
The purpose of this trial is to study the effect of Human Papillomavirus (HPV) vaccination on the elevation of antibody titer to 4 serotypes of HPV in patients with systemic lupus erythematous and compare the antibody response with an equal number of age-matched healthy women.

DETAILED DESCRIPTION:
Genital infection with human papillomavirus (HPV) is one of the most common sexually transmitted infections in Hong Kong. Most cases of HPV infection are asymptomatic. However, in some individuals, especially those patients who are immunocompromised, HPV infection is persistent and may result in genital warts, cervical smear abnormalities, cervical intraepithelial neoplasia (CIN) and rarely cervical cancer.

Systemic lupus erythematosus (SLE) is a disease that predominantly affects women of the childbearing age. Patients with SLE are at risk of persistent HPV infection. This is because of the immunosuppressive state induced by various treatments. The prevalence of abnormal Pap smears and cervical squamous intraepithelial neoplasia (CIN) in SLE patients is higher than that in age-matched healthy women. Thus, prevention of HPV infection is important in patients with SLE to reduce the incidence of CIN lesions and hence invasive cervical cancers in the long run.

The quadrivalent HPV vaccine, GARDASIL is effective in reducing the occurrence of high-grade CIN lesions and anogenital disease elated to HPV-16 and HPV-18 infection. Vaccination of young women aged 16 to 23 years resulted in seroconversion rates of more than 99% for all the HPV types (6,11,16,18) and was well tolerated. There has been very little information regarding the efficacy of the quadrivalent HPV vaccine in immunocompromised hosts. The objectives of the current study are to evaluate the immunogenicity and safety of the quadrivalent HPV vaccine in a group of patients with SLE in terms of antibody conversion. Comparison will be made with an equal number of age-matched healthy women.

ELIGIBILITY:
Inclusion Criteria:

SLE patients

* Female patients aged ≤ 35 years
* Fulfilling the American College of Rheumatology (ACR) criteria for the classification of SLE
* Having received a stable dose of prednisolone and/or other immunosuppressive agents within 3 months of study entry
* Able to give written informed consent

Controls

* Women aged ≤ 35 years, matched those of SLE patients recruited
* No known chronic medical diseases
* Not receiving any long-term medications including herbs

Exclusion Criteria:

* History of allergy to HPV vaccines

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
antibody titers against 4 strains of human papillomavirus | baseline, month 7 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital, Hong Kong, China
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Ho LY, To CH. Long-term immunogenicity of a quadrivalent human papillomavirus vaccine in systemic lupus erythematosus. Vaccine. 2018 May 31;36(23):3301-3307. doi: 10.1016/j.vaccine.2018.04.056. Epub 2018 Apr 24. PMID 29699792